CLINICAL TRIAL: NCT01856816
Title: Effect of Meal Patterning on Carotenoid Absorption From Vegetables
Acronym: S26
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Purdue University (Other)
Responsible Party: Principal Investigator, Wayne Campbell, Prof. Foods and Nutrition, Purdue University
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: 1102010527
Record Dates: First submitted 2013-05-15; First posted 2013-05-17 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2013-05

CONDITIONS: Carotenoid; Bioavailability; Dietary Modification

STUDY DESIGN:
Who Masked: Investigator

ARMS (3):
- Meal Pattern Treatment A (Experimental): A large vegetable salad (262g) and with a moderate amount of canola oil (8g) was consumed over a two meal period as designated by treatment group A.
  Interventions: Other: Meal Pattern Treatment A
- Meal Pattern Treatment B (Experimental): A large vegetable salad (262g) and with a moderate amount of canola oil (8g) was consumed over a two meal period as designated by treatment group B.
  Interventions: Other: Meal Pattern Treatment B
- Treatment Group C (Other): A large vegetable salad (262g) and with a moderate amount of canola oil (8g) was consumed over a two meal period as designated by treatment group C.
  Interventions: Other: Meal Pattern Treatment C

INTERVENTIONS:
Other: Meal Pattern Treatment A — In treatment A, subjects consumed 100% of salad vegetables and canola oil in the first meal and 0% in the second. Additional protein-rich "chef's salad" ingredients were distributed equally between meals.
  Arms: Meal Pattern Treatment A
Other: Meal Pattern Treatment B — In treatment B, subjects consumed 50% of salad vegetables and canola oil in the first meal and 50% in the second. Additional protein-rich "chef's salad" ingredients were distributed equally between meals.
  Arms: Meal Pattern Treatment B
Other: Meal Pattern Treatment C — In treatment C, subjects consumed 75% of vegetables and oil in the first meal and 25% in the second. Additional protein-rich "chef's salad" ingredients were distributed equally between meals.
  Arms: Treatment Group C

SUMMARY:
The purpose of this research study is to determine how different meal patterns influence the absorption of beneficial plant pigments (carotenoids) from vegetables. The hypothesis is that carotenoid absorption will be lower when daily vegetables are consumed in one meal compared two smaller meals throughout the day.

ELIGIBILITY:
Inclusion criteria:

* Age range: 18-50 years
* Body mass index (BMI: weight (kg)/height (m2)) ranging from 20-29 kg/m²
* Weight stable (<4.5 kg change within the last 3 months)
* Constant habitual activity pattern, not to exceed activities of a recreational level over the past 3 months
* Have clinically normal blood profiles (specifically normal liver and kidney functions and fasting blood glucose of ≤110 mg/dl)
* Non-smoking
* Non-diabetic
* No current use of medication affecting lipid profile
* No intestinal disorders including lipid malabsorption, lactose intolerance
* No heavy consumption of alcohol (>2 drinks per day)
* No current use of dietary supplements that affect cholesterol, (e.g. Benocol or fiber supplements) or a willingness to discontinue their use during the study

Exclusion criteria:

* Diabetic
* Use of lipid altering medications

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2011-05; Primary Completion 2011-07 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Area under the concentration (AUC) vs time curve for carotenoids in the triglyceride-rich lipoprotein (TRL) fraction of plasma. | 0, 2, 3, 4, 5, 6, 7, 8, 9, 10, 12 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Mario Ferruzzi, PhD, Principal Investigator — Purdue University; Wayne Campbell, PhD, Principal Investigator — Purdue University